CLINICAL TRIAL: NCT03248219
Title: Sleep Disordered Breathing Accounts for Abnormal Glycemic Profiles in Pregnant Women: The Sleep in Pregnancy (SiP) Study
Brief Title: The Sleep in Pregnancy Study
Acronym: SiP
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado Clinical & Translational Sciences Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 16-2568
Record Dates: First submitted 2017-08-07; First posted 2017-08-14 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Pregnancy Related; Sleep Disordered Breathing; Obesity
MeSH Terms: conditions — Sleep Apnea Syndromes; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sleep disordered breathing (SDB) insidiously worsens metabolic function, heightens insulin resistance (IR), and in pregnancy is thought to precipitate gestational diabetes, preterm birth, growth restriction, gestational hypertension, and preeclampsia. Despite the fact that sleep disturbances are common during pregnancy, SDB remains under-recognized, under-diagnosed, and poorly understood, particularly in pregnancies affected by obesity. Sixty percent of pregnancies are now affected by obesity, yet the relationship between SDB, patterns of glycemia, and insulin resistance (IR) in obese pregnant women is a neglected area with major therapeutic implications to improve maternal and infant health. Using a prospective design in which diet and gestational age are highly controlled, the investigators propose to measure SDB (apneas/hypopneas) in obese pregnant women using an ambulatory sleep monitoring system. In parallel, robust patterns of glycemia will be measured with a continuous glucose monitoring system (CGMS), followed by a 75g oral glucose tolerance test to measure insulin action. The investigators global hypothesis is that worse SDB in part accounts for higher 24-hour patterns of glycemia in obese normal glucose tolerant (NGT) pregnant women in their 3rd trimester. The Investigators will test the hypothesis that: 1) In obese NGT pregnant women at 32-34 weeks gestation on a controlled eucaloric diet, higher apnea hypopnea index (AHI) will be positively associated with 24-hour glycemia measured by a CGMS and that, 2) Higher AHI in obese NGT pregnant women at 32-34 weeks gestation on a eucaloric controlled diet will be associated with higher insulin resistance measured by a 75g oral glucose tolerance test (Matsuda Model). Early identification and treatment has the potential to decrease long-term maternal cardiovascular morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women:

  1. Between the ages of 20-39 yrs,
  2. At 32-34 weeks gestation,
  3. Who have a BMI of ≥30 to ≤40 kg/m2,
  4. Who have a singleton pregnancy, and
  5. Who have a normal glucose tolerance test on entrance to the study.

Exclusion Criteria:

* Pregnant Women:

  1. Who have a diagnosis of diabetes (GDM, type 1 or type 2),
  2. Who are using beta blockers/glucocorticoids.
  3. Who have other children who are ≤2 yrs old (due to risk of disrupted sleep),
  4. With diagnosed sleep disorders (e.g. OSA, insomnia, restless leg syndrome),
  5. Who work night or rotating shifts,
  6. Who report use of sleep medications will be excluded,
  7. With diagnosed pulmonary or cardiovascular disease
  8. Who do not speak English.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women who are 32-34 weeks pregnant who live in the Denver Metro Area
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
24 hour glycemia measurement of the Pregnant Mother | Every 24 hours for 3 days
  Glycemia will be measured by Continuous glucose monitoring
Evaluation of Insulin resistance of the Pregnant Mother | 2 hours after a 75 gram glucose load
  Insulin resistance will be measured with an Oral Glucose Tolerance Test

SECONDARY OUTCOMES:
Infant Body Composition | At 2 weeks of life
  Percent of Fat Mass
Stress Levels | 15 minutes before Sleep and 15 minutes after sleep
  Cortisol Levels

CONTACTS AND LOCATIONS:
Overall Officials: Sarah S Farabi, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No